CLINICAL TRIAL: NCT01563731
Title: European Society of Hypertension and Chinese Hypertension League Stroke in Hypertension Optimal Treatment Trial
Brief Title: Optimal Blood Pressure and Cholesterol Targets for Preventing Recurrent Stroke in Hypertensives
Acronym: ESH-CHL-SHOT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Collaborators: European Society of Hypertension (Other); Chinese Hypertension League (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 27F201
Record Dates: First submitted 2012-03-20; First posted 2012-03-27 (Estimated); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Stroke; Transient Ischemic Attack; Hypertension
Keywords: Blood pressure medicines; Lipid lowering medicines; Hypertension; Stroke; Dementia; Heart attack; Heart failure
MeSH Terms: conditions — Stroke; Ischemic Attack, Transient; Hypertension; Dementia; Myocardial Infarction; Heart Failure | interventions — Calcium Channel Blockers; Angiotensin-Converting Enzyme Inhibitors; Angiotensin Receptor Antagonists; Sodium Chloride Symporter Inhibitors; Adrenergic beta-Antagonists; Adrenergic alpha-Antagonists; Mineralocorticoid Receptor Antagonists; Simvastatin; Pravastatin; Fluvastatin; Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- SBP < 145-135 mmHg and LDL-C 2.8 - 1.8 mmol/l (Other): Highest SBP target. Higher LDL-C target. Control arm
  Interventions: Drug: all approved antihypertensive drugs; all approved statins
- SBP < 135-125 mmHg and LDL-C 2.8 - 1.8 mmol/l (Active Comparator): Intermediate SBP target. Higher LDL-C target
  .
  Interventions: Drug: all approved antihypertensive drugs; all approved statins
- SBP < 125 mmHg and LDL-C 2.8 - 1.8 mmol/l (Active Comparator): Lowest SBP target. Higher LDL-C target
  Interventions: Drug: all approved antihypertensive drugs; all approved statins
- SBP < 145-135 mmHg and LDL-C < 1.8 mmol/l (Active Comparator): Highest SBP target. Lower LDL-C target.
  Interventions: Drug: all approved antihypertensive drugs; all approved statins
- SBP < 135-125 mmHg and LDL-C < 1.8 mmol/l (Active Comparator): Intermediate SBP target. Lower LDL-C target.
  Interventions: Drug: all approved antihypertensive drugs; all approved statins
- SBP < 125 mmHg and LDL-C < 1.8 mmol/l (Active Comparator): Lowest SBP target. Lower LDL-C target.
  Interventions: Drug: all approved antihypertensive drugs; all approved statins

INTERVENTIONS:
Drug: all approved antihypertensive drugs; all approved statins — All drugs to be used at doses capable of bringing SBP and LDL-C to targets; only doses approved in each country.
  Other Names: Calcium channel blockers; Angiotensin converting enzyme inhibitors; Angiotensin receptor blockers; Thiazide diuretics; Beta-blockers; Alpha-blockers; Aldosterone antagonists; Simvastatin; Pravastatin; Fluvastatin; Atorvastatin; Rosuvastatin

SUMMARY:
Stroke is one of the major causes not only of mortality, but of disease burden worldwide, because of residual disability and cognitive decline. Although blood pressure lowering has been clearly shown to be the most effective means for primary and secondary prevention of stroke, the systolic blood pressure (SBP) levels to achieve by treatment in order to optimize prevention results are unknown, and whether SBP levels lower than those usually recommended are accompanied by further or reduced benefits is undecided yet. Likewise, while low-density lipoprotein cholesterol (LDL-C) lowering by statins has been shown to be associated with primary and secondary stroke prevention, whether more intense lowering is or is not of further benefit is unknown. The Stroke in Hypertension Optimal Treatment Trial (ESH-CHL-SHOT) is a factorial 3 x 2 arm, multicenter, randomized clinical trial designed to test the hypothesis that in elderly patients at high risk of recurrent stroke (previous recent stroke or TIA) antihypertensive treatment programs aimed at reducing SBP to the usually recommended values (< 145 to 135 mmHg), to a lower goal (< 135 to 125 mmHg) or to even lower values (< 125 mmHg) will result in progressively greater reductions in recurrent stroke, incidence of cardiovascular outcomes and cognitive decline. Parallely, the preventive efficacy of more and less intense LDL-C reductions will be tested on the same outcomes.

DETAILED DESCRIPTION:
ESH-CHL-SHOT will randomize about 7500 participants aged > or = 65 years with SBP > or = 140 mmHg or antihypertensive therapy, who have presented a stroke or TIA, within 1 to 6 months before randomization.

The trial will investigate

1. the effects of randomization to antihypertensive treatment of different intensities, aiming at three different SBP targets. SBP targets are < 145 to 135, < 135 to 125, < 125 mmHg, with approximate mean inter-target differences of 8 mmHg;
2. the effects of randomization to lipid lowering treatment of different intensity, aiming at two different LDL-C targets. Targets are 2.8 to 1.8 mmol/l (110 to 70 mg/dl) and < 1.8 mmol/l;
3. possible interactions between antihypertensive and lipid-lowering treatments. The primary hypothesis is that recurrent stroke rates will be 25% lower in the lowest vs intermediate SBP target group, 25% lower in the intermediate vs higher SBP target group, and 20% lower in the lower vs higher LDL-C target group. Sample size has been calculated to provide a 80% power with a significance of 5% after corrections for repetitive measurements on the assumption that stroke incidence will be 4% per year in the highest SBP target group. Participants will be recruited at approximately 250 clinics in Europe (2500 patients) and China (5000 patients) over a 2-year period, and will be followed up for an average of 4 years or until 925 recurrent strokes occur.

Arms and assigned intervention

1. Antihypertensive treatment design and assigned treatment

Participants will be randomly allocated to one of three different sitting SBP targets:

1. < 145 to 135 mmHg
2. < 135 to 125 mmHg
3. < 125 mmHg to be possibly achieved within 3 months and subsequently maintained within the target window.

Investigators are free to choose the drugs (among those approved in each country) to be administered to individual patients. It is expected that patients already on antihypertensive therapy and with SBP at randomization not too far from target will be maintained on current therapy with suitable adjustments. Other patients (untreated or with SBP far from target) may follow a suggested treatment algorithm of progressive increase in number of compounds or doses. During follow-up visits drugs and/or doses will be modified if necessary to maintain patients within randomized target window.

2. Lipid-lowering treatment design and assigned treatment

Participants will be randomly allocated to one of two different LDL-C targets:

A) 2.8 to 1.8 mmol/l (110 to 70 mg/dl) B) < 1.8 mmol/l (< 70 mg/dl) to be possibly achieved within 3 months and subsequently maintained within the target window.

Investigators are free to choose the statin (among those approved in each country) to be administered to individual patients. The initial statin dose should be chosen by the investigator according to LDL-C at randomization and the LDL-C target. The initial dose can be increased (to the maximum dose allowed in each country) or decreased until the LDL-C target is achieved possibly within 3 months, and further adjusted up or down at 6-month intervals in order to maintain LDL-C within the randomized target window.

ELIGIBILITY:
Inclusion Criteria:

* Qualifying event: stroke or TIA 1 to 6 months previous to randomization.
* All patients should have a CT scan or MRI (preferably MRI) at screening. The CT scan or MRI carried out at the time of the qualifying event, if available, is acceptable. Stroke will be defined as imaging evidence of a recent brain infarction (or haemorrhage) independently of duration of clinical symptoms, or as duration of clinical symptoms > 24 h even in absence of imaging evidence of lesion
* TIA as clinical symptoms (involving limbs or speech) lasting < 24 h without imaging evidence of infarction. Enrolling units should avoid enrolling patients with TIA in a proportion greater than 25% of enrolled patients. The general coordinators in Milan and Beijing may decide stopping enrolment of TIA patients if their proportion is becoming greater than expected.
* A haemorrhagic stroke (1 to 6 months previously) is also a qualifying event, but only for the BP-lowering component of the trial (see Exclusion criteria).
* Age: 65 years and above. No fixed upper age limit is introduced, but frail patients aged above 80 years should not be enrolled.
* Gender: either gender.
* BP: Only hypertensive patients: untreated patients with SBP ≥140 mmHg; patients on antihypertensive treatment with any BP (but see exclusion criteria)
* LDL-C: Patients without statin treatment with LDL-C > 2.8 mmol/l; patients on statin treatment with any LDL-C value (but see exclusion criteria)
* Antiplatelet therapy: All patients should be under antiplatelet therapy (agents and doses chosen by the investigator according to accepted guidelines), unless contraindicated. Anticoagulant (instead of antiplatelet) therapy whenever indicated (e.g. atrial fibrillation).

Exclusion Criteria:

* Qualifying event:

  1. Patients in unstable clinical conditions
  2. Clinical disturbances caused by non-stroke pathology
  3. patients with haemodynamically significant carotid stenosis or requiring carotid revascularization
  4. haemorrhagic stroke is an exclusion criterion for the lipid lowering component of the trial; however, these patients should be randomized to the BP component, but considered in addition to the number of patients requested to each enrolling unit, in order not to decrease the power of the lipid-lowering component.
* BP: - known secondary hypertension;
* SBP >140 mmHg under three antihypertensive drugs at full doses (these patients are unlikely to achieve SBP < 125 mmHg, if so randomized);
* orthostatic hypotension (SBP fall > 25 mmHg on standing);
* LDL-C: - LDL-C >2.8 mmol/l under full dose of a statin (these patients are unlikely to achieve LDL-C targets).
* LDL-C > 4.5 mmol/l under low dose of a statin or untreated (these patients are unlikely to achieve the lower LDL-C target).
* Others: - Patients with a myocardial infarction (preceding or subsequent to the qualifying stroke or TIA) if their baseline LDL-C is < 1.8 mmol/l
* Dementia
* Severe disability (modified Rankin scale > 4)
* Severe chronic renal failure defined as serum creatinine > 250 micromol/l
* Hepatic disease as determined by either AST or ALT values > 2 times the upper limit of normal
* History of hepatic encephalopathy, esophageal varices or portocaval shunt
* History of gastrointestinal surgery or disorders which could interfere with drug absorption
* Known allergy or contraindications to one of the drugs to be administered in the study
* History of malignancy including leukaemia and lymphoma (but not basal cell skin cancer) within the last 5 years
* History of clinically significant autoimmune disorders such as systemic lupus erythematosus
* History of drug or alcohol abuse within the last 5 years
* History of non-compliance to medical regimens and/or patients who are considered potentially unreliable
* Inability or unwillingness to give free informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Recurrent stroke | five years
  Time to occurrence of (recurrent) stroke (fatal and non fatal)

SECONDARY OUTCOMES:
Major cardiovascular (CV) events | five years
  First major cardiovascular events, a composite of CV death, non fatal stroke, non fatal myocardial infarction, vascular intervention, hospitalized heart failure
Cognitive impairment and dementia | five years
  Cognitive impairment (decline in Montreal Cognitive Assessment Test); Dementia (Disability Assessment for Dementia)

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Zanchetti, Principal Investigator — Istituto Auxologico Italiano; Lisheng Liu, MD, Principal Investigator — Beijing Hypertension League Institute
Locations (1):
- Almazov Federal Heart, Blood and Endocrinology Centre, Saint Petersburg, Russia

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623
- [Derived] Zanchetti A, Liu L, Mancia G, Parati G, Grassi G, Stramba-Badiale M, Silani V, Bilo G, Corrao G, Zambon A, Scotti L, Zhang X, Wang H, Zhang Y, Zhang X, Guan TR, Berge E, Redon J, Narkiewicz K, Dominiczak A, Nilsson P, Viigimaa M, Laurent S, Agabiti-Rosei E, Wu Z, Zhu D, Rodicio JL, Ruilope LM, Martell-Claros N, Pinto F, Schmieder RE, Burnier M, Banach M, Cifkova R, Farsang C, Konradi A, Lazareva I, Sirenko Y, Dorobantu M, Postadzhiyan A, Accetto R, Jelakovic B, Lovic D, Manolis AJ, Stylianou P, Erdine S, Dicker D, Wei G, Xu C, Xie H, Coca A, O'Brien J, Ford G. Blood pressure and LDL-cholesterol targets for prevention of recurrent strokes and cognitive decline in the hypertensive patient: design of the European Society of Hypertension-Chinese Hypertension League Stroke in Hypertension Optimal Treatment randomized trial. J Hypertens. 2014 Sep;32(9):1888-97. doi: 10.1097/HJH.0000000000000254. PMID 24979303